#### **Protocol C3991009**

A PHASE 1, OPEN-LABEL, SINGLE-DOSE, PARALLEL GROUP STUDY TO COMPARE THE PHARMACOKINETICS OF PF-07081532 IN ADULT PARTICIPANTS WITH VARYING DEGREES OF HEPATIC IMPAIRMENT RELATIVE TO PARTICIPANTS WITHOUT HEPATIC IMPAIRMENT

Statistical Analysis Plan (SAP)

Version: 1

**Date:** 10Aug-2022

## TABLE OF CONTENTS

| LIST OF TABLES | .3 |
|---|---|
| LIST OF FIGURES | .4 |
| APPENDICES | 4 |
| 1. VERSION HISTORY | 5 |
| 2. INTRODUCTION | 5 |
| 2.1. Modifications to the Analysis Plan Described in the Protocol | 5 |
| 2.2. Study Objectives, Endpoints, and Estimands | 5 |
| 2.2.1. Primary Estimand(s) | 6 |
| 2.2.2. Secondary Estimand(s) | 6 |
| 2.2.3. Additional Estimand(s) | 6 |
| 2.3. Study Design | 6 |
| 3. ENDPOINTS AND BASELINE VARIABLES: DEFINITIONS AND CONVENTIONS | 7 |
| 3.1. Primary Endpoint(s) | 7 |
| 3.2. Secondary Endpoint(s) | 8 |
| CCI | |
| 3.4. Baseline Variables | 9 |
| 3.5. Safety Endpoints | C |
| 4. ANALYSIS SETS (POPULATIONS FOR ANALYSIS) | 0 |
| 5. GENERAL METHODOLOGY AND CONVENTIONS | 0 |
| 5.1. Hypotheses and Decision Rules | 1 |
| 5.2. General Methods | 1 |
| 5.2.1. Analyses for Continuous Endpoints | 1 |
| 5.2.2. Analyses for Categorical Endpoints | 1 |
| 5.2.3. One-way Analysis of Variance (ANOVA) | 1 |
| 5.2.4. Linear Regression PK Parameters versus Hepatic Function | 1 |
| CCI | |
| 5.3. Methods to Manage Missing Data | 2 |
| 5.3.1. Pharmacokinetic Concentrations Below the Limit of Quantification 1 | |

| 5.3.3. Pharmacokinetic Parameters 13 6. ANALYSES AND SUMMARIES 13 6.1. Primary Endpoint(s) 13 6.1.1. PF-07081532 PK Parameters 13 6.1.1.1. Main Analysis 13 6.1.1.2. Sensitivity/Supplementary Analyses 14 6.2. Secondary Endpoint(s) 14 6.2.1. Adverse Events 15 6.2.2. Laboratory Data 15 6.2.3. Vital Signs 15 6.2.4. ECG 15 CCI CCI 6.4. Subset Analyses 17 6.5. Baseline and Other Summaries and Analyses 17 6.5.1. Baseline Summaries 17 6.5.2. Study Conduct and Participant Disposition 17 6.5.3. Study Treatment Exposure 17 6.5.4. Concomitant Medications and Nondrug Treatments 17 6.6. Safety Summaries and Analyses 18 7.1. Introduction 18 7.2. Interim Analyses and Summaries 18 8. REFERENCES 18 APPENDICES 19 | | . Pharmacokinetic Deviations, Missing Concentrations and nomalous Values | 13 |
|---|---|---|---|
| 6. ANALYSES AND SUMMARIES 13 6.1. Primary Endpoint(s) 13 6.1.1. PF-07081532 PK Parameters 13 6.1.1. Main Analysis 13 6.1.1. Main Analysis 14 6.2. Secondary Endpoint(s) 14 6.2. Secondary Endpoint(s) 15 6.2.1. Adverse Events 15 6.2.2. Laboratory Data 15 6.2.3. Vital Signs 15 6.2.4. ECG 15 6.5. Baseline and Other Summaries and Analyses 17 6.5.1. Baseline Summaries 17 6.5.2. Study Conduct and Participant Disposition 17 6.5.3. Study Treatment Exposure 17 6.5.4. Concomitant Medications and Nondrug Treatments 17 6.6. Safety Summaries and Analyses 18 7. INTERIM ANALYSES 18 7.1. Introduction 18 7.2. Interim Analyses and Summaries 18 8. REFERENCES 18 APPENDICES 19 | | | |
| 6.1. Primary Endpoint(s) | 6. ANALYSES A | AND SUMMARIES | 13 |
| 6.1.1. PF-07081532 PK Parameters | | | |
| 6.1.1.2. Sensitivity/Supplementary Analyses 14 6.2. Secondary Endpoint(s) 14 6.2.1. Adverse Events 15 6.2.2. Laboratory Data 15 6.2.3. Vital Signs 15 6.2.4. ECG 15 6.1 15 6.2.1. Baseline and Other Summaries and Analyses 17 6.5.1. Baseline Summaries 17 6.5.2. Study Conduct and Participant Disposition 17 6.5.3. Study Treatment Exposure 17 6.6. Safety Summaries and Analyses 18 7. INTERIM ANALYSES 18 7.1. Introduction 18 7.2. Interim Analyses and Summaries 18 8. REFERENCES 18 APPENDICES 19 | | | |
| 6.2. Secondary Endpoint(s) 14 6.2.1. Adverse Events 15 6.2.2. Laboratory Data 15 6.2.3. Vital Signs 15 6.2.4. ECG 15 SCI 6.4. Subset Analyses 17 6.5. Baseline and Other Summaries and Analyses 17 6.5.1. Baseline Summaries 17 6.5.2. Study Conduct and Participant Disposition 17 6.5.3. Study Treatment Exposure 17 6.5.4. Concomitant Medications and Nondrug Treatments 17 6.6. Safety Summaries and Analyses 18 7. INTERIM ANALYSES 18 7.1. Introduction 18 7.2. Interim Analyses and Summaries 18 8. REFERENCES 18 APPENDICES 19 | | 6.1.1.1. Main Analysis | 13 |
| 6.2. Secondary Endpoint(s) 14 6.2.1. Adverse Events 15 6.2.2. Laboratory Data 15 6.2.3. Vital Signs 15 6.2.4. ECG 15 SCI 6.4. Subset Analyses 17 6.5. Baseline and Other Summaries and Analyses 17 6.5.1. Baseline Summaries 17 6.5.2. Study Conduct and Participant Disposition 17 6.5.3. Study Treatment Exposure 17 6.5.4. Concomitant Medications and Nondrug Treatments 17 6.6. Safety Summaries and Analyses 18 7. INTERIM ANALYSES 18 7.1. Introduction 18 7.2. Interim Analyses and Summaries 18 8. REFERENCES 18 APPENDICES 19 | | • | |
| 6.2.2. Laboratory Data 15 6.2.3. Vital Signs 15 6.2.4. ECG 15 SGI 6.4. Subset Analyses 17 6.5. Baseline and Other Summaries and Analyses 17 6.5.1. Baseline Summaries 17 6.5.2. Study Conduct and Participant Disposition 17 6.5.3. Study Treatment Exposure 17 6.5.4. Concomitant Medications and Nondrug Treatments 17 6.6. Safety Summaries and Analyses 18 7. INTERIM ANALYSES 18 7.1. Introduction 18 7.2. Interim Analyses and Summaries 18 8. REFERENCES 18 APPENDICES 19 | 6.2. Second | | |
| 6.2.3. Vital Signs 15 6.2.4. ECG 15 SCI 6.4. Subset Analyses 17 6.5. Baseline and Other Summaries and Analyses 17 6.5.1. Baseline Summaries 17 6.5.2. Study Conduct and Participant Disposition 17 6.5.3. Study Treatment Exposure 17 6.5.4. Concomitant Medications and Nondrug Treatments 17 6.6. Safety Summaries and Analyses 18 7. INTERIM ANALYSES 18 7.1. Introduction 18 7.2. Interim Analyses and Summaries 18 8. REFERENCES 18 APPENDICES 19 | 6.2.1. | Adverse Events | 15 |
| 6.2.4. ECG 15 6.6.1. Subset Analyses 17 6.5. Baseline and Other Summaries and Analyses 17 6.5.1. Baseline Summaries 17 6.5.2. Study Conduct and Participant Disposition 17 6.5.3. Study Treatment Exposure 17 6.5.4. Concomitant Medications and Nondrug Treatments 17 6.6. Safety Summaries and Analyses 18 7. INTERIM ANALYSES 18 7.1. Introduction 18 7.2. Interim Analyses and Summaries 18 8. REFERENCES 18 APPENDICES 19 | 6.2.2. | Laboratory Data | 15 |
| 6.4. Subset Analyses | 6.2.3. | Vital Signs | 15 |
| 6.4. Subset Analyses 17 6.5. Baseline and Other Summaries and Analyses 17 6.5.1. Baseline Summaries 17 6.5.2. Study Conduct and Participant Disposition 17 6.5.3. Study Treatment Exposure 17 6.5.4. Concomitant Medications and Nondrug Treatments 17 6.6. Safety Summaries and Analyses 18 7. INTERIM ANALYSES 18 7.1. Introduction 18 7.2. Interim Analyses and Summaries 18 8. REFERENCES 18 APPENDICES 19 | 6.2.4. | ECG | 15 |
| 6.5. Baseline and Other Summaries and Analyses 17 6.5.1. Baseline Summaries 17 6.5.2. Study Conduct and Participant Disposition 17 6.5.3. Study Treatment Exposure 17 6.5.4. Concomitant Medications and Nondrug Treatments 17 6.6. Safety Summaries and Analyses 18 7. INTERIM ANALYSES 18 7.1. Introduction 18 7.2. Interim Analyses and Summaries 18 8. REFERENCES 18 APPENDICES 19 | CCI | | |
| 6.5. Baseline and Other Summaries and Analyses 17 6.5.1. Baseline Summaries 17 6.5.2. Study Conduct and Participant Disposition 17 6.5.3. Study Treatment Exposure 17 6.5.4. Concomitant Medications and Nondrug Treatments 17 6.6. Safety Summaries and Analyses 18 7. INTERIM ANALYSES 18 7.1. Introduction 18 7.2. Interim Analyses and Summaries 18 8. REFERENCES 18 APPENDICES 19 | | | |
| 6.5. Baseline and Other Summaries and Analyses 17 6.5.1. Baseline Summaries 17 6.5.2. Study Conduct and Participant Disposition 17 6.5.3. Study Treatment Exposure 17 6.5.4. Concomitant Medications and Nondrug Treatments 17 6.6. Safety Summaries and Analyses 18 7. INTERIM ANALYSES 18 7.1. Introduction 18 7.2. Interim Analyses and Summaries 18 8. REFERENCES 18 APPENDICES 19 | | | |
| 6.5. Baseline and Other Summaries and Analyses 17 6.5.1. Baseline Summaries 17 6.5.2. Study Conduct and Participant Disposition 17 6.5.3. Study Treatment Exposure 17 6.5.4. Concomitant Medications and Nondrug Treatments 17 6.6. Safety Summaries and Analyses 18 7. INTERIM ANALYSES 18 7.1. Introduction 18 7.2. Interim Analyses and Summaries 18 8. REFERENCES 18 APPENDICES 19 | | | |
| 6.5. Baseline and Other Summaries and Analyses 17 6.5.1. Baseline Summaries 17 6.5.2. Study Conduct and Participant Disposition 17 6.5.3. Study Treatment Exposure 17 6.5.4. Concomitant Medications and Nondrug Treatments 17 6.6. Safety Summaries and Analyses 18 7. INTERIM ANALYSES 18 7.1. Introduction 18 7.2. Interim Analyses and Summaries 18 8. REFERENCES 18 APPENDICES 19 | 64.61.4 | A 1 | 17 |
| 6.5.1. Baseline Summaries | | | |
| 6.5.2. Study Conduct and Participant Disposition 17 6.5.3. Study Treatment Exposure 17 6.5.4. Concomitant Medications and Nondrug Treatments 17 6.6. Safety Summaries and Analyses 18 7. INTERIM ANALYSES 18 7.1. Introduction 18 7.2. Interim Analyses and Summaries 18 8. REFERENCES 18 APPENDICES 19 | | | |
| 6.5.3. Study Treatment Exposure 17 6.5.4. Concomitant Medications and Nondrug Treatments 17 6.6. Safety Summaries and Analyses 18 7. INTERIM ANALYSES 18 7.1. Introduction 18 7.2. Interim Analyses and Summaries 18 8. REFERENCES 18 APPENDICES 19 | | | |
| 6.5.4. Concomitant Medications and Nondrug Treatments | | | |
| 6.6. Safety Summaries and Analyses | | | |
| 7. INTERIM ANALYSES | | _ | |
| 7.1. Introduction | _ | - | |
| 7.2. Interim Analyses and Summaries | | | |
| 8. REFERENCES | | | |
| APPENDICES19 | | | |
| LIST OF TABLES | THE LINDICES | | 1) |
| | | LIST OF TABLES | |
| Table 1. Summary of Changes | Table 1. | Summary of Changes | 5 |

| Table 2. | Hepatic Function Categories Based on Child-Pugh Score6 |
|---|---|
| | y of Plasma PK Parameters of PF-07081532 to be calculated |
| | y of Plasma PK parameters of Unbound PF-07081532 to be calculated8 |
| CCI | |
| | y statistics to be produced for Plasma PK Parameters of PF-0708153214 |
| CCI | |
| | LIST OF FIGURES |
| No table of figur | es entries found. |
| | APPENDICES |
| Table 1. | Summary of Changes5 |
| Table 2. | Hepatic Function Categories Based on Child-Pugh Score6 |
| Table 3. Summar | y of Plasma PK Parameters of PF-07081532 to be calculated7 |
| Table 4. Summar | y of Plasma PK parameters of Unbound PF-07081532 to be calculated8 |
| CCI | |
| Table 7. Summar | y statistics to be produced for Plasma PK Parameters of PF-0708153214 |
| CCI | |
| Appendix 1. Stati | stical Methodology Details |
| Appendix 2. Cate | gorical Classes for ECG and Vital Signs of Potential Clinical Concern20 |
| Appendix 3. List | of Abbreviations21 |

#### 1. VERSION HISTORY

Table 1. Summary of Changes

| Version/<br>Date | Associated<br>Protocol<br>Amendment | Rationale | Specific Changes |
|---|---|---|---|
| 1<br>10 AUG2022 | Original<br>18 May 2022 | N/A | N/A |

#### 2. INTRODUCTION

PF-07081532 is an oral GLP-1R agonist that is currently being investigated as a chronic therapy to improve glycemic control in adult participants with T2DM. Based on review of the effect of hepatic impairment on human PK for compounds cleared in a similar manner to PF-07081532 (OATP-mediated hepatic uptake), impaired hepatic function is generally associated with increased drug exposures in plasma.

Therefore, the primary purpose of this study is to characterize the effect of varying degrees of hepatic impairment on the plasma PK of PF-07081532 following administration of a single oral dose of PF-07081532.

This statistical analysis plan (SAP) provides the detailed methodology for summary and statistical analyses of the data collected in Study C3991009.

#### 2.1. Modifications to the Analysis Plan Described in the Protocol

Not Applicable

#### 2.2. Study Objectives, Endpoints, and Estimands

| Objectives | Endpoints |
|---|---|
| Primary: | Primary: |
| To compare the PK of PF-07081532 following administration of a single oral dose in adult participants with varying degrees of hepatic impairment relative to age- and body weight-matched participants without hepatic impairment. | • Plasma: C <sub>max</sub> , AUC <sub>inf</sub> , AUC <sub>last</sub> *, fu, C <sub>max,u</sub> , AUC <sub>inf,u</sub> and AUC <sub>last,u</sub> *, as data permit. |
| Secondary: | Secondary: |
| To evaluate the safety and tolerability of a single oral dose of PF-07081532 when administered to adult participants with varying degrees of hepatic impairment and in age- and body weight-matched participants without hepatic impairment. | Assessment of treatment emergent AEs, clinical laboratory abnormalities, vital signs, ECG parameters. |
| CCI | |



\*  $AUC_{last}$  and  $AUC_{last,u}$  will be treated as primary endpoints if data do not permit robust estimation of  $AUC_{inf}$  and  $AUC_{inf,u}$ 

#### 2.2.1. Primary Estimand(s)

Not applicable because C3991009 is a Phase 1 study with no estimands on PK endpoints

#### 2.2.2. Secondary Estimand(s)

Not applicable because C3991009 is a Phase 1 study with no estimands on safety endpoints

## 2.2.3. Additional Estimand(s)

Not applicable because C3991009 is a Phase 1 study with no estimands on safety endpoints

#### 2.3. Study Design

This is an open-label, single-dose, parallel-group, multicenter study to investigate the effect of varying degrees of hepatic function on the plasma PK of PF-07081532 after a single, oral 20 mg dose administered in the fed state (standard breakfast). Safety and tolerability will be evaluated throughout the study. A total of approximately 24 participants with varying degrees of hepatic function will be dosed in the study as shown in Table 2. If recruitment of participants with severe hepatic impairment proves prohibitive, the number of participants to be enrolled in this group may be flexible (4-6 participants).

Table 2. Hepatic Function Categories Based on Child-Pugh Score

| Group | Description | Child-Pugh Score | Number of Participants |
|---|---|---|---|
| 1 | Without hepatic impairment | Not Applicable | $6^a$ |
| 2 | Mild hepatic impairment | Class A (5 to 6 points) | 6 |
| 3 | Moderate hepatic impairment | Class B (7 to 9 points) | 6 |
| 4 | Severe hepatic impairment | Class C (10 to 15 points) | $6^b$ |

a. Additional participants may be dosed to a maximum of 8 participants to ensure mean age  $\pm 5$  years and mean body weight  $\pm 10$  kg of this group is aligned with the pooled averageassessed when approximately  $\geq 75\%$  of participants are dosed across the other 3 groups.

Categorization of participants into Groups 2-4 will be done based on Child-Pugh scores determined at the screening visit, as described in Appendix 11 of the protocol.

b. If recruitment proves to be prohibitive, study may dose 4-6 participants in this group.

## Staged Enrollment of Study Groups

Participants will be dosed in a staged manner as follows:

- Participants with moderate and severe hepatic impairment (Groups 3 and 4) will be enrolled first.
- Recruitment of participants with mild hepatic impairment (Group 2) will initiate when approximately 50% of the participants across Groups 3 and 4 have been dosed.

## Sponsor approval is required <u>before</u> proceeding with recruitment of Group 2.

- An average value for age and weight for the 3 hepatic impairment groups (Groups 2-4) will be determined, and participants without hepatic impairment (Group 1) will be recruited to match the average demographics (at a minimum, age and weight, and as much as practically possible gender) across the pooled Groups 2-4.
- Recruitment for healthy participants in Group 1 (without hepatic impairment) may start when approximately 75% of total participants across Groups 2-4 (ie, approximately 12-13 participants) have been dosed.

Sponsor approval is required before proceeding with recruitment of Group 1.

# 3. ENDPOINTS AND BASELINE VARIABLES: DEFINITIONS AND CONVENTIONS

Baseline is defined as the last pre-dose assessment for all endpoints, unless otherwise specified.

#### 3.1. Primary Endpoint(s)

• PF-07081532 Plasma Pharmacokinetic parameters: C<sub>max</sub>, AUC<sub>inf</sub>, AUC<sub>last</sub>, fu, C<sub>max,u</sub>, AUC<sub>inf,u</sub>, AUC<sub>last,u</sub> as data permit.

The plasma PK parameters in Table 3 will be derived from concentration-time profiles using standard non-compartmental analysis methods (with the exception of fu that will be directly determined by the analytical lab):

Table 3. Summary of Plasma PK Parameters of PF-07081532 to be calculated

| Parameter | Analysis<br>Scale | PF-07081532 20mg |
|----------------------|-------------------|------------------|
| $C_{max}$ | ln | A, D |
| AUC <sub>inf</sub> * | ln | A, D |
| $AUC_{last}^+$ | ln | A, D |
| fu | R | A, D |
| $C_{max,u}$ | ln | A, D |

| AUC <sub>inf,u</sub> * | ln | A, D |
|------------------------|----|------|
| $AUC_{last,u}^+$ | ln | A, D |

<sup>\*=</sup>if data permits. +AUC<sub>last</sub> and AUC<sub>last,u</sub> will be treated as primary endpoints if data do not permit robust estimation of AUC<sub>inf</sub> and AUC<sub>inf,u</sub>,

Abbreviations: A = analyzed using a statistical model; D=displayed with descriptive statistics as outlined in Table 7 in Section 6.1.1.1; ln=natural-log transformed; R=raw (untransformed).

The plasma PK parameters for unbound PF-07081532 will be calculated as described in Table 4:

Table 4. Summary of Plasma PK parameters of Unbound PF-07081532 to be calculated

| Parameter | Method of Determination |
|------------------------|---------------------------|
| $AUC_{last,u}^+$ | $fu \times AUC_{last}$ |
| AUC <sub>inf,u</sub> * | fu × AUC <sub>inf</sub> * |
| $C_{max,u}$ | $fu \times C_{max}$ |

<sup>\*=</sup>if data permits. <sup>+</sup>AUC<sub>last</sub> and AUC<sub>last,u</sub> will be treated as primary endpoints if data do not permit robust estimation of AUC<sub>inf</sub> and AUC<sub>inf,u</sub>,

#### 3.2. Secondary Endpoint(s)

Assessment of treatment emergent AEs, clinical laboratory abnormalities, vital signs, ECG parameters.

An adverse event is considered treatment emergent (TEAE) relative to a given treatment if:

• the event starts during the effective duration of treatment (i.e. starting on or after the dose of PF-07081532 but before this dose plus lag time)

The effective duration of treatment is determined by the lag time. Any event occurring within the lag time is attributed to the corresponding treatment. The lag time is defined by the Pfizer Standard of 365 days post last dose of IP.

A 3-tier approach for summarizing AEs will not be used due to the low number of participants planned to be recruited.

The following data are considered in standard safety summaries (see protocol for collection days and list of parameters):

- adverse events,
- laboratory data,
- vital signs data,
- ECG results.

For laboratory, vital signs and ECG data, baseline will be defined as the last pre-dose measurement, unless otherwise specified.



#### 3.4. Baseline Variables

Not Applicable.

#### 3.5. Safety Endpoints

See Section 3.2

## 4. ANALYSIS SETS (POPULATIONS FOR ANALYSIS)

Data for all participants will be assessed to determine if participants meet the criteria for inclusion in each analysis population prior to unblinding and releasing the database and classifications will be documented per standard operating procedures.

For purposes of analysis, the following analysis sets are defined:

| Participant Analysis Set | Description |
|---|---|
| Enrolled | "Enrolled" means a participant's, or their legally authorized representative's, agreement to participate in a clinical study following completion of the informed consent process and assignment to study intervention. A participant will be considered enrolled if the informed consent is not withdrawn prior to participating in any study activity after screening. Potential participants who are screened for the purpose of determining eligibility for the study, but do not participate in the study, are not considered enrolled, unless otherwise specified by the protocol. |
| Safety analysis set | All participants assigned to study intervention and who take at least 1 dose of study intervention. |
| PK Concentration Set | The PK concentration population is defined as all participants who received at least 1 dose of PF-07081532 and in whom at least 1 plasma concentration value is reported. |
| PK Parameter Set | The PK parameter analysis population is defined as all participants who received at least 1 dose of PF-07081532 and have at least 1 of the PK parameters of interest calculated. |
| CCI | |

#### 5. GENERAL METHODOLOGY AND CONVENTIONS

The following group labels (or similar) will be used for tables and figures unless otherwise stated:

| Group | Description of Group | Label |
|-------|-----------------------------|-----------------------------|
| 1 | Normal hepatic function | Without Hepatic Impairment |
| 2 | Mild hepatic impairment | Mild Hepatic Impairment |
| 3 | Moderate hepatic impairment | Moderate Hepatic Impairment |
| 4 | Severe hepatic impairment | Severe Hepatic Impairment |

#### 5.1. Hypotheses and Decision Rules

There is no statistical hypothesis testing planned for this study and no statistical decision rules will be applied.

#### 5.2. General Methods

#### 5.2.1. Analyses for Continuous Endpoints

Unless otherwise stated, continuous endpoints and relevant safety endpoints will be presented using summary statistics: number of observations, arithmetic mean, standard deviation, median, minimum and maximum values.

#### 5.2.2. Analyses for Categorical Endpoints

Categorical endpoints and relevant safety endpoints will be presented using summary statistics: number of observations, counts and percentages.

#### 5.2.3. One-way Analysis of Variance (ANOVA)

The one-way analysis of variance (ANOVA) model will include group as a factor.

Estimates of the adjusted mean differences (Test - Reference), and corresponding 90% CIs, will be obtained from the model. These will be exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios. Example SAS code is given in Appendix 1.

Residuals from the models will be examined for normality and the presence of outliers via visual inspection of plots of residuals vs predicted values and normal probability plots of residuals but these will not be included in the clinical study report. If there are major deviations from normality or outliers (where studentized residuals are greater than 3 or less than - 3) then the effect of these on the conclusions may be investigated through alternative transformations and/or analyses excluding outliers. Justification for any alternative to the planned analysis will be given in the report of the study if applicable.



#### 5.2.4. Linear Regression PK Parameters versus Hepatic Function

Linear regression will be used to analyze the potential relationship between appropriate PK parameters (eg, AUC<sub>inf</sub>, AUC<sub>last</sub>, C<sub>max</sub>, fu, AUC<sub>inf</sub>, AUC<sub>last</sub>, C<sub>max</sub>, fu, AUC<sub>inf</sub>, AUC<sub>last</sub>, C<sub>max</sub>, and hepatic function as a continuous explanatory variable (using either continuous serum albumin, prothrombin time or total bilirubin, each modelled separately). Estimates of the slope and intercept, together

with a 90% CI, and the coefficient of determination (i.e. R-squared and adj-R-squared) may be obtained from the model. Example SAS code is given in Appendix 1.

Residuals from the models will be examined for normality and the presence of outliers via visual inspection of plots of residuals vs predicted values and normal probability plots of residuals but these will not be included in the clinical study report. If there are major deviations from normality or outliers (where studentized residuals are greater than 3 or less than - 3) then the effect of these on the conclusions may be investigated through alternative transformations and/or analyses excluding outliers. Alternative model structure may also be considered. Justification for any alternative to the planned analysis will be given in the report of the study if applicable.



#### 5.3. Methods to Manage Missing Data

For the analysis of safety endpoints, the sponsor data standard rules for imputation will be applied.

#### 5.3.1. Pharmacokinetic Concentrations Below the Limit of Quantification

In all data presentations (except listings), concentrations below the limit of quantification (BLQ) will be set to zero. In listings BLQ values will be reported as "<LLQ", where LLQ will be replaced with the value for the lower limit of quantification.

#### 5.3.2. Pharmacokinetic Deviations, Missing Concentrations and Anomalous Values

In summary tables and plots of median/mean profiles, statistics will be calculated having set concentrations to missing if 1 of the following cases is true:

- 1. A concentration has been collected as ND (ie, not done) or NS (ie, no sample),
- 2. A deviation in sampling time is of sufficient concern or a concentration has been flagged anomalous by the pharmacokineticist/clinical team.

Note that summary statistics will not be presented at a particular time point if more than 50% of the data are missing.

#### 5.3.3. Pharmacokinetic Parameters

Actual PK sampling times will be used in the derivation of PK parameters.

If a PK parameter cannot be derived from a participant's concentration data, the parameter will be coded as NC (ie, not calculated). Note that NC values will not be generated beyond the day that a participant discontinues.

In analysis and summary tables, statistics will be calculated by setting NC values to missing; and statistics will be presented for a particular group with  $\geq 3$  evaluable measurements.

If an individual participant has a known biased estimate of a PK parameter (due for example to an unexpected event such as vomiting before all the compound is adequately absorbed in the body), this will be footnoted in summary tables/figures and will not be included in the calculation of summary statistics or statistical analyses.

#### 6. ANALYSES AND SUMMARIES

Data collected before baseline will only be listed, unless otherwise stated.

Unless otherwise stated, all analyses, summaries and listings will be produced by group (as outlined in Section 5) which would include all 4 groups in the same analysis/output.

#### 6.1. Primary Endpoint(s)

#### 6.1.1. PF-07081532 PK Parameters

• Estimand strategy: Not applicable

• Analysis set: PF-07081532 Concentration and Pharmacokinetic Parameter Set

#### 6.1.1.1. Main Analysis

C<sub>max</sub>, AUC<sub>inf</sub> (if data permit), AUC<sub>last</sub>, fu, AUC<sub>inf,u</sub>, AUC<sub>last,u</sub> and C<sub>max,u</sub> will be listed, summarized descriptively and analyzed by group for participants in the PK parameter set (as defined in Section 4). Missing values will be handled as detailed in Section 5.3.

A one-way analysis of variance (ANOVA) described in Section 5.2.3, that includes all 4 groups in the same model, will be used to compare the natural log transformed of  $C_{max}$ ,  $AUC_{inf}$ ,  $AUC_{inf}$ ,  $AUC_{inf,u}$ ,  $AUC_{inf,u}$ ,  $AUC_{inf,u}$ , and  $C_{max,u}$  of PF-07081532 separately, for each of the hepatic impairment groups (Test, Groups 2, 3, 4) to the healthy normal hepatic function group (Reference, Group 1).

For summary statistics and median or mean plots by sampling time, the nominal PK sampling time will be used. For individual participant plots by time, the actual PK sampling time will be used. The plasma PK parameters of PF-07081532 for each group will be summarized as specified in Table 7 below.

Table 7. Summary statistics to be produced for Plasma PK Parameters of PF-07081532

| Parameter | Summary Statistics |
|---|---|
| C <sub>max</sub> , AUC <sub>inf</sub> *, AUC <sub>last</sub> , fu, | N, arithmetic mean, median, cv%, standard deviation, |
| AUCinf,u*, AUClast,u, and | minimum, maximum, geometric mean and geometric |
| $C_{\text{max,u}}$ | cv%. |

<sup>\*</sup> if data permits

The following plots will be presented:

• Box and whisker plots for individual PK parameters ( $AUC_{inf}$ ,  $AUC_{last}$ ,  $C_{max}$ ,  $f_u$ ,  $AUC_{inf,u}$ ,  $AUC_{last,u}$  and  $C_{max,u}$ )) will be constructed by group and overlaid with geometric means.

#### 6.1.1.2. Sensitivity/Supplementary Analyses



Plots of PK parameters (eg, AUC<sub>inf</sub>, AUC<sub>last</sub>, C<sub>max</sub>, f<sub>u</sub>, AUC<sub>inf</sub>, AUC<sub>last</sub>, and C<sub>max</sub>, u) versus hepatic function at baseline (e.g. serum albumin, prothrombin time or total bilirubin, plotted separately) will be constructed, with a regression line and 90% confidence region included from the main linear regression model.

#### 6.2. Secondary Endpoint(s)

Any clinical laboratory, ECG, BP, and pulse rate abnormalities of potential clinical concern will be described.

No formal analyses are planned for safety data.

The safety endpoints detailed in Section 3.2 will be listed and summarized in accordance with sponsor reporting standards based on the safety population (as defined in Section 4), with more details provided below.

#### **6.2.1.** Adverse Events

Adverse events will be summarised by group and overall, in accordance with sponsor reporting standards using the safety population defined in Section 4.

If applicable, subject discontinuations due to adverse events will be detailed and summarized.

#### 6.2.2. Laboratory Data

Laboratory data will be listed and summarized by group and overall, in accordance with the sponsor reporting standards using the safety population defined in Section 4. Baseline is as defined in Section 3.2.

#### 6.2.3. Vital Signs

Absolute values and changes from baseline in seated systolic and diastolic blood pressure and pulse rate will be summarised by group, according to sponsor reporting standards using the safety population defined in Section 4. Baseline is as defined in Section 3.2.

Maximum and minimum absolute values and maximum changes from baseline for seated vital signs will also be summarised descriptively by group using categories as defined in Appendix 2. Numbers and percentages of participants meeting the categorical criteria will be provided. All planned and unplanned post dose time points will be counted in these categorical summaries. All values meeting the criteria of potential clinical concern will be listed.

#### 6.2.4. ECG

Absolute values and changes from baseline in QT interval, heart rate, QTcF interval, PR interval and QRS interval will be summarised by group using sponsor reporting standards and the safety population defined in Section 4. Tables will be paged by parameter. Baseline is as defined in Section 3.2.

Maximum absolute values and changes from baseline for QTcF, PR and QRS will also be summarised descriptively by group using categories as defined in Appendix 2. Numbers and percentages of participants meeting the categorical criteria will be provided. All planned and unplanned post dose time points will be counted in these categorical summaries. All values meeting the criteria of potential clinical concern will be listed.







#### 6.4. Subset Analyses

No subset analyses will be performed.

## 6.5. Baseline and Other Summaries and Analyses

Data will be reported in accordance with the sponsor reporting standards.

#### **6.5.1.** Baseline Summaries

Demographics data (age, biological sex, race, ethnicity, weight, body mass index and height) will be summarized by group and overall, as outlined in Sections 5.2.1 and 5.2.2 as applicable.

#### 6.5.2. Study Conduct and Participant Disposition

Participant evaluation groups will show end of study participant disposition by group and will show which participants were analyzed for pharmacokinetics and safety, which may not be produced in one table. Frequency counts and percentages will be supplied for participant discontinuation(s) by group.

#### 6.5.3. Study Treatment Exposure

Not applicable.

#### 6.5.4. Concomitant Medications and Nondrug Treatments

All prior and concomitant medication(s) as well as non-drug treatment(s) will be provided in listings.

#### 6.6. Safety Summaries and Analyses

See Section 6.2.

#### 7. INTERIM ANALYSES

#### 7.1. Introduction

No formal interim analysis will be conducted for this study. As this is an open-label study, the sponsor may conduct unblinded reviews of the data during the course of the study for the purpose of safety assessment, facilitating PK modeling, and/or supporting clinical development.

## 7.2. Interim Analyses and Summaries

Not applicable.

#### 8. REFERENCES

None.

#### **APPENDICES**

## **Appendix 1. Statistical Methodology Details**

```
An example of SAS code for ANOVA:
proc mixed data = tab.pk;
       class group;
       model l&var = group /residual;
       lsmeans group/diff cl alpha=0.1;
       ods output lsmeans = lsmeans&var;
       ods output diffs=diffs&var;
run;
An example of SAS code for the PROC REG code for linear regression analyses:
proc reg data=tab.pk;
       model l&var=clcr/clb alpha=0.1;
       ods output ParameterEstimates = param&var;
       ods output FitStatistics = fit&var;
       ods output ANOVA = reg\&var;
run;
An example of SAS code for stepwise regression with model selection using AIC:
proc glmselect data=tab.pk analysis plot=ALL;
  model pk p = albumin age weight/ selection=stepwise (select = AIC stop = AIC)
       include=1 hierarchy=none showpvalues;
run;
```

## Appendix 2. Categorical Classes for ECG and Vital Signs of Potential Clinical Concern Categories for QTcF

| Absolute value of QTcF (msec) | >450 and ≤480 | >480 and ≤500 | >500 |
|---------------------------------------|---------------|---------------|------|
| Increase from baseline in QTcF (msec) | >30 and ≤60 | >60 | |

## **Categories for PR and QRS**

| PR (ms) | max. ≥300 | |
|---|---|---|
| PR (ms) increa se from baseline | | Baseline ≤200 and max.≥50% increase |
| QRS (ms) | max. ≥140 | |
| QRS (ms) increase from baseline | ≥50% increase | |

## **Categories for Vital Signs**

| Systolic BP (mm Hg) | min. <90 | |
|---|---|---|
| Systolic BP (mm Hg) change from baseline | max. decrease ≥30 | max. increase ≥30 |
| Diastolic BP (mm Hg) | min. <50 | |
| Diastolic BP (mm Hg) change from baseline | max. decrease ≥20 | max. increase ≥20 |
| Seatedpulse rate (bpm) | min. <40 | max. >120 |

Measurements that fulfill these criteria are to be listed in the report.

## Appendix 3. List of Abbreviations

| Abbreviation | Term |
|------------------|-----------------------------------|
| AE | adverse event |
| Ae | Amount excreted |
| ANOVA | analysis of variance |
| AUC | area under the curve |
| BLQ | below the limit of quantitation |
| BP | blood pressure |
| CI | confidence interval |
| CL | Clearance |
| CCI | |
| $C_{\text{max}}$ | maximum observed concentration |
| CCI | |
| CSR | clinical study report |
| CV | Coefficient of variation |
| ECG | Electrocardiogram |
| IP | Investigational Product |
| LLQ | Lower limit of quantitation |
| Ln | Natural log |
| N/A | not applicable |
| NC | not calculated |
| ND | not done |
| NS | no sample |
| PK | pharmacokinetic(s) |
| QTc | corrected QT |
| QTcF | corrected QT (Fridericia method) |
| SAP | statistical analysis plan |
| SOA | Schedule of activities |
| TEAE | Treatment emergent adverse events |
| CCI | |